CLINICAL TRIAL: NCT04648566
Title: Endometrium Immunomodulation Using in Utero Administration of Peripheral Blood Mononuclear Cells
Brief Title: Endometrium Immunomodulation by in Utero Administration of Peripheral Blood Mononuclear Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fertilys (Industry)
Collaborators: Institut National de la Recherche Scientifique - Centre Armand Frappier Santé Biotechnologie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Immunomodulation
Record Dates: First submitted 2020-11-18; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IIU control group (Placebo Comparator)
  Interventions: Procedure: Intrauterine administration of sperm washing medium
- IIU PBMC group (Active Comparator)
  Interventions: Procedure: Intrauterine administration of hCG-activated peripheral blood mononuclear cells
- FIV control group (Placebo Comparator)
  Interventions: Procedure: Intrauterine administration of sperm washing medium
- FIV PBMC group (Active Comparator)
  Interventions: Procedure: Intrauterine administration of hCG-activated peripheral blood mononuclear cells
- RIF group (Active Comparator)
  Interventions: Procedure: Intrauterine administration of hCG-activated peripheral blood mononuclear cells

INTERVENTIONS:
Procedure: Intrauterine administration of hCG-activated peripheral blood mononuclear cells — Administration of hCG-activated peripheral blood mononuclear cells in the uterine cavity of the patient
  Arms: FIV PBMC group; IIU PBMC group; RIF group
Procedure: Intrauterine administration of sperm washing medium — Administration of sperm washing medium instead of PBMC in the uterine cavity of the patient
  Arms: FIV control group; IIU control group

SUMMARY:
One of the most limiting factors in the field of assisted reproduction is implantation failure. A new approach to increase the chances of success involves the use of cells from the patient's blood, peripheral blood mononuclear cells (PBMC), which once isolated can be cultured for a few days and then inseminated back into the uterine cavity prior to embryo implantation. It has been shown that the immune system plays a major role in the process of embryo implantation. To date, at least three international clinical trials appear to confirm the usefulness of intrauterine administration of PBMC in the setting of repeated implantation failure (RIF) in in vitro fertilization (IVF) (RIF: absence of active pregnancy after ≥ 3 embryo transfers). The clinical pregnancy rate would be doubled or even tripled. This treatment has never been studied in a randomized double-blind clinical trial, in the context of fertilization without RIF or in a classic treatment such as intrauterine insemination (IUI) with the partner sperm.

Our hypothesis is that the creation of an endometrial inflammatory reaction by the administration of PBMC in the uterine cavity allows a better receptivity and consequently a better implantation following an embryo transfer as part of an IVF treatment.

The objective is to evaluate whether intrauterine administration of PBMC improves embryo implantation following assisted reproduction treatment.

The investigators plan to recruit 148 women undergoing IVF and 220 patients undergoing UII with partner sperm to test our hypothesis. The investigators also plan to recruit all RIF patients accepting to participate in the clinical trial. The study will be prospective, randomized and double-blind. The treated group will receive an intrauterine administration of PBMC while the control group will be administered with sperm washing medium only. PBMC will be obtained from a blood sample (maximum 10 ml) a few days before embryo transfer in IVF cases or on the day of sperm insemination in IUI cases. PBMC will then be isolated in the laboratory on a Ficoll gradient in order to eliminate platelets, polynuclear cells and red blood cells. PBMCs will then be stimulated with phytohemagglutinin (PHA) and human chorionic gonadotropin hormone (hCG) for 48 hours. Lymphocyte phenotyping will be assessed before and after cell activation. In addition, the cytokine profile will be established from the supernatant of the stimulated cells. These data will make it possible to establish a link between the pro-versus anti-inflammatory cytokine profile and implantation success versus failure for each patient. Two days after cell seeding, PBMC will be administered into the uterine cavity of the patient. Embryo transfer will be performed in the same way as the standard treatment on day 3 or 5 according to the criteria established by the IVF laboratory and in agreement with the doctor.

ELIGIBILITY:
Inclusion Criteria:

* All infertile patients undergoing in vitro fertilization (IVF) or intrauterine insemination (IUI) with partner's sperm at Fertilys, agreeing to participate in the study and having signed the study participation consent form.
* Study participants must be over 18 years old.
* For the recurrent implantation failure (RIF) group only: Patients described as having RIF, i.e. having had ≥ 3 good quality embryo transfers.

Exclusion Criteria:

* For the randomized IUI and IVF groups only: Patients described as having RIF, i.e. having had ≥ 3 embryo transfers or having had a transfer of more than 3 embryos of good quality.
* Patients requiring a donation of gametes (eggs or spermatozoa).
* Couples in which one or the other has a chromosomal abnormality.
* Patients who are starting an IUI cycle under ovulation testing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Biochemical pregnancy rate | Two weeks following embryo transfer or 3 weeks following intrauterine insemination
Clinical pregnancy rate | Six to 8 weeks of gestation

SECONDARY OUTCOMES:
Peripheral blood mononuclear cells populations distribution at Day 0 | The day of the patient's ovulation
Peripheral blood mononuclear cells populations distribution at Day 2 | After 48 hours of culture
Cytokines expression levels | After 48 hours of culture

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Miron, MD, PhD, Principal Investigator — Fertilys inc
Locations (1):
- Fertilys inc., Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No